CLINICAL TRIAL: NCT06347367
Title: Investigation of Short-term Effect of Exercise and Self-manual Approaches to Core Muscles Patients With Bloating - Distention
Brief Title: Short-term Effect of Exercise and Self-manual Approaches to Bloating - Distention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gulruh Karabagli, Master degree student of physiotherapy and rehabilitation, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EU-FTR-GK-01
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Gastrointestinal System Disease; Functional Bloating; Distension; Bowel; Gastrointestinal Motility Disorder; Pelvic Floor Dyssynergia
Keywords: Functional bloating; distension; gastrointestinal motility; exercise therapy; pelvic floor
MeSH Terms: conditions — Digestive System Diseases; Dilatation, Pathologic | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to Group 1 (exercise and self-manual approaches targeting only the diaphragm muscles) and Group 2 (exercise and self-manual approaches targeting both diaphragm and core muscles).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator and Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (exercise and self-manual approaches targeting only the diaphragm muscles) (Active Comparator): Diaphragmatic stretching technique, pectoral muscle relaxation, diaphragmatic mobilisation, thoracic mobilisation and diaphragmatic breathing.
  Interventions: Other: Group 1 (exercise and self-manual approaches targeting only the diaphragm muscles)
- Group 2 (exercise and self-manual approaches targeting both diaphragm and core muscles) (Active Comparator): İn addition to Group 1, patients in group 2 will receive, abdominal massage, abdominal mobilisation, stabilisation exercises and pelvic floor muscle training.
  Interventions: Other: Group 2 (exercise and self-manual approaches targeting both diaphragm and core muscles)

INTERVENTIONS:
Other: Group 1 (exercise and self-manual approaches targeting only the diaphragm muscles) — Both groups will receive the patient education before treatment. Diaphragmatic stretching technique, pectoral muscle relaxation, diaphragmatic mobilisation, thoracic mobilisation and diaphragmatic breathing. Exercise and self-manual approaches will be performed at home 3 times a day for 8 repetitions for 4 weeks and approximately 45-60 minutes.
  Arms: Group 1 (exercise and self-manual approaches targeting only the diaphragm muscles)
Other: Group 2 (exercise and self-manual approaches targeting both diaphragm and core muscles) — İn addition to Group 1, patients in group 2 will receive, abdominal massage, abdominal mobilisation, stabilisation exercises and pelvic floor muscle training. Exercise and self-manual approaches will be performed at home 3 times a day for 8 repetitions for 4 weeks and approximately 45-60 minutes.
  Arms: Group 2 (exercise and self-manual approaches targeting both diaphragm and core muscles)

SUMMARY:
Abdominal bloating and distension (ABD) are the most commonly gastrointestinal symptoms reported by patients with various functional gut disorders such as functional dyspepsia, irritable bowel syndrome and it is frequently associated with constipation. The pathophysiology of ABD is complex, often multifactorial and poorly understood. The reseach was hypothesised that short-term self-manual approaches and exercise for core muscles would have a positive effect on the symptoms of ABD.

DETAILED DESCRIPTION:
Characteristic symptoms include recurrent abdominal fullness, pressure, or a sensation of trapped gas (abdominal bloating), and/or measurable increase in abdominal girth (abdominal distention). There are several key components in pathophysiology of ABD: a subjective sensation of abdominal bloating, objective abdominal distention, volume of intra-abdominal contents, altered pelvic floor muscle function and muscular activity of the abdominal wall. Therapeutic options include; dietary modifications, probiotics, antibiotics, prokinetic agents, antispasmodics, neuromodulators, biofeedback and physical activity. However, treatment of ABD is limited and not effective in all individuals with this symptom. There is no study investigated the effectiveness of exercise and self-manual approaches in patients with ABD. Therefore, investigators aim to determine the short-term effects and differences of exercise and self-manual approaches on symptoms in patients with ABD. Women between the ages of 18 and 75 who meet the Rome Ⅳ criteria will be diagnosed with ABD by Ege University Faculty of Medicine, Department of Gastroenterology will be included in the study. Participants will be assigned to Group 1 (exercise and self-manual approaches targeting only the diaphragm muscles) and Group 2 (exercise and self-manual approaches targeting both diaphragm and core muscles). Exercise and self-manual approaches will be performed at home 3 times a day for 8 repetitions for 4 weeks and approximately 45-60 minutes. Both groups will receive the patient education before treatment. Group 1 exercise and self-manual program include; diaphragmatic stretching technique, pectoral muscle relaxation, diaphragmatic mobilisation, thoracic mobilisation and diaphragmatic breathing. İn addition to Group 1, patients in group 2 will receive, abdominal massage, abdominal mobilisation, stabilisation exercises and pelvic floor muscle training. ABD symptoms will be assessed on a 6-point graphic rating scale (Perception of sensations), Gastrointestinal Symptom Rating Scale (GSRS), Diaphragm, abdominal wall and pelvic floor muscle and other related muscles will be assessed with Surface Electromyography (SEMG), High-Resolution Anorectal Manometry (HRAM), Balloon Expulsion Test (BET), Colon transit time (CTT) and Ultrasonography (USG).

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages of 18 and 75
* Diagnosed with abdominal bloating-distension according to the Rome IV criteria
* Without any condition preventing exercise
* Proficiency in Turkish reading and writing

Exclusion Criteria:

* Individuals with any organic cause for bloating and distension (such as celiac disease or other absorption disorders, intestinal dysmotility, and chronic intestinal pseudo-obstruction)
* Those with alarm symptoms (weight loss, rectal bleeding, or anemia)
* A history of major gastrointestinal or abdomino-pelvic surgery
* Who unable to complete the study protocol
* Cognitively challenged to the extent that it would hinder the conduct of the study
* Pregnant individuals

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females between the ages of 18 and 75 who meet the Rome Ⅳ criteria will be diagnosed with ABD
Enrollment: 24 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-17 (Estimated); Study Completion 2024-06-19 (Estimated)

PRIMARY OUTCOMES:
Abdominal bloating and distention (ABD) Perception of sensations | Pre-intervention; immediately after the Four weeks
  A graded questionnaire will be used to measure the intensity and the type of sensations perceived, and an anatomical questionnaire to measure the location and extension of the perceived sensations. The graded questionnaire included four sensations: pressure, fullness, colicky sensation, and stinging sensation. Each sensation will independently scored on a graphic rating scale that combined verbal descriptors on a visual analogue scale graded from 0 to 6 (0 represent no Perception at all, score 5 represent discomfort, and score 6 represent a painful sensation). The anatomic questionnaire will be showed the abdomen divided in nine areas corresponding to epigastrium, periumbilical area, hypogastrium, both hypochondria, flanks, and ileal fossae, and the participants were instructed to mark the location, abdominal area(s) or extra-abdominal, where the sensations were perceived. Before the study, both questionnaires will be fully explained to the participants.

SECONDARY OUTCOMES:
Superficial Electromyography (EMG) | Pre-intervention; immediately after the Four weeks
  A NeuroTrac MyoPlus 4 PRO (Verity Medical, UK) type EMG device will be used in the study. Bioelectrical activities of the muscles (pelvic floor muscles, abdominal muscles, diaphragm, multifidus) will be recorded with disposable 3.2 x 3.2 cm superficial electrodes. To reduce skin impedance, the skin area will be cleaned with an alcohol swab. Active electrodes will be placed on the right side of the body, parallel to the muscle fibers, according to the reference points. The reference electrode will be placed on the anterior superior iliac spine. Measurements will be performed during six seconds of maximal voluntary contraction ('work' phase EMG activity) and six seconds of relaxation ('rest' phase EMG activity) of the pelvic floor muscles. Measurements will be repeated for three times. The graphic and numerical data provided by the device will be recorded in the evaluation form.

OTHER OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS) | Pre-intervention; immediately after the Four weeks
  It is a Likert-type scale with 15 items developed to assess symptoms related to gastrointestinal disorders, ranging from 'no discomfort' to 'very severe discomfort.' The scale's 15 items consist of five subscales: abdominal pain, reflux, diarrhea, indigestion, and constipation. Questions 1, 4, and 5 assess abdominal pain; questions 2 and 3 assess reflux; questions 11, 12, and 14 assess diarrhea; questions 6, 7, 8, and 9 assess indigestion; and questions 10, 13, and 15 assess constipation, and the evaluation is made accordingly. High scores obtained from the GSRS indicate more severe symptoms.
High-resolution anorectal manometry (HRAM) | Pre-intervention; immediately after the Four weeks
  To evaluate recto-anal reflex activity, anal sphincter function, recto-anal coordination during simulated defecation, and rectal sensory function will be utilized Medical Measurement Systems (MMS) device (Model- SOLAR SYSTEM, 771459). HRAM assessment will be conducted according to the London Classification. The evaluation will involve placing an air-charged (UniTip High Resolution Catheter (Unisensor)) lubricated manometry probe, equipped with pressure sensors, gently into the rectum while the patient is in the left lateral position, with the most distal sensor (1 cm level) positioned posteriorly 1 cm from the anal verge. Subsequently, approximately 3 minutes will be allotted for the patient to return to baseline anal tone. Anal resting pressure, short squeeze pressure, endurance squeeze pressure, cough reflex, push pressure, Recto-Anal İnhibitory Reflex (RAIR), rectal sensation will be evaluated.
Balloon Expulsion Test (BET) | Pre-intervention; immediately after the Four weeks
  After completing the anorectal manometry test, the Balloon Expulsion Test (BET) will be conducted by inserting an Anorectal Reflex Balloon Catheter (ADS) into the rectum, with a non-latex balloon lubricated with gel measuring 4-5 cm in length. Subsequently, the patient will be provided with privacy. While in a seated position, the balloon will be filled with 50 ml of warm water, and the patient will be asked to sit on a commode chair and expel the balloon. The patient will be instructed to start the timer, begin straining, and stop the timer when the balloon is expelled. Healthy individuals typically can expel a 50 ml balloon in less than 1 minute. Duration shorter than 2 minutes will be considered normal.
Colon Transit Time (CTT) | Pre-intervention; immediately after the Four weeks
  Colon Transit Time (CTT) will provide a quantitative assessment of colonic motor function. Participants in both groups will be instructed to ingest 10 radio-opaque ring-shaped markers (Transit-Pellets, Medifactia, Stockholm, Sweden) consecutively for 5 days each morning at 09:00. On the 6th day, they will be asked to ingest 5 stick-shaped markers at 09:00 and the remaining 5 at 21:00 (to measure rapid transit). Approximately 12 hours after the last marker intake (144 hours in total on Day 7), abdominal radiographs will be taken. The retained markers will be counted for the ascending colon, transverse colon, descending colon, sigmoid colon, and rectum. If the number of retained markers is less than 5, it will be analyzed as normal colonic transit.
Ultrasonography (USG) | Pre-intervention; immediately after the Four weeks
  The ultrasound assessment will be conducted using a Siemens X700 device equipped with a 2-dimensional, 3.5- megahertz transducer in B mode, both transabdominally and transperineally with a curvilinear probe. Prior to measurement, a standard bladder filling protocol will be employed. Measurements including diaphragm, intercostal muscles, upper and lower rectus abdominis, external and internal oblique abdominals, transversus abdominis, multifidus, erector spinae, and rectus diastasis will be recorded in millimeters (mm). Additionally, measurements of the anorectal angle and anopubic angle will be recorded in degrees (°). Measurements will be taken during inspiration, expiration, and pelvic floor contraction.
Digital dynamometer | Pre-intervention; immediately after the Four weeks
  A digital dynamometer (handheld dynamometer (HHD)) will be utilized to determine trunk flexor and extensor muscles isometric strength. Measurements will be recorded as the average of two maximum repetitions following warm-up. Results will be documented in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Nuray ELİBOL, Study Director — Ege University; Gülruh KARABAĞLI, Principal Investigator — Ege University; Melahat AKTAŞ, Principal Investigator — Dokuz Eylul University; Özge ÇELİKER TOSUN, Principal Investigator — Dokuz Eylul University; Serhat BOR, Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Medicine, Department of Gastroenterology, Izmir, Bornova, Turkey (Türkiye)